CLINICAL TRIAL: NCT03105882
Title: Pilot Study of Clinical Safety and Feasibility of the Neuro-Spinal Scaffold for the Treatment of Complete (AIS A) Traumatic Acute Spinal Cord Injury at the C5 - T1 Neurological Levels
Brief Title: Pilot Study of the Neuro-Spinal Scaffold for the Treatment of AIS A Cervical Acute SCI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not enroll any subjects.
Sponsor: InVivo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: InVivo-100-102
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Traumatic Cervical Acute Spinal Cord Injury
Keywords: Spinal Cord Injury; SCI; Complete (AIS A) Traumatic Acute Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neuro-Spinal Scaffold (Experimental)
  Interventions: Device: Neuro-Spinal Scaffold

INTERVENTIONS:
Device: Neuro-Spinal Scaffold — Experimental: Neuro-Spinal Scaffold

SUMMARY:
Pilot Study of Clinical Safety and Feasibility of the Neuro-Spinal ScaffoldTM for the Treatment of Complete (AIS A) Traumatic Acute Spinal Cord Injury at the C5-T1 Neurological Levels The purpose of this study is to support an expansion to support marketing applications as well as future studies.

ELIGIBILITY:
Inclusion Criteria:

* 16-70 years of age, inclusive
* AIS A classification of traumatic spinal cord injury with a neurological level within C5-T1 inclusive
* Recent injury
* Non-penetrating SCI

Exclusion Criteria:

* Terminally ill subjects not likely to be able to participate in follow-up
* Incomplete spinal cord injury (AIS B, C, D, and E injuries)
* No identifiable intra-spinal cavity following myelotomy/irrigation in the contused spinal cord in which a Scaffold can be placed
* Spinal cord injury associated with significant traumatic brain injury or coma that
* Radiographic or visual evidence of parenchymal dissociation or anatomic transection as determined by the Investigator where the contusion completely bridges a full cross-section of the spinal cord
* Subjects with spinal cord injuries directly due to gunshot, knife, or other penetrating wounds

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of all Adverse Device Effects of any kind/seriousness. | 6 Months

OTHER OUTCOMES:
American Spinal Injury Association Impairment Scale (AIS) improvement of one or more grade | 6 months
  International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Exams
Improvements in motor and sensory scores | 6 months
  ISNCSCI exams
Improvements in Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) | 6 months
  GRASSP Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Toselli, MD, Study Director — InVivo Therapeutics
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada